CLINICAL TRIAL: NCT07013292
Title: Retrospective Bicentric Study in a Cohort of French Friedreich's Ataxia Patients on the 6-month Efficacy of Omaveloxolone Treatment on Dysphagia.
Brief Title: Efficacy of Omaveloxolone Treatment for Dysphagia in French Patients With Friedreich's Ataxia
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Neuro02
Record Dates: First submitted 2025-05-23; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — omaveloxolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Friedreich ataxia treated with Omaveloxolone: SKYCLARYS (omaveloxolone)
  Interventions: Drug: SKYCLARYS (omaveloxolone)

INTERVENTIONS:
Drug: SKYCLARYS (omaveloxolone) — Skyclarys is indicated for the treatment of Friedreich's ataxia in adults and adolescents aged 16 and over. Opaque capsule with "RTA 408" printed in white ink on the light green body and "50" printed in white ink on the blue cap. Capsules (size 0) measure 21.7 ± 0.3 mm in length and the outer diameter of the cap is 7.64 ± 0.06 mm. Omaveloxolone should be initiated and monitored by physicians experienced in treating patients with patients with Friedreich's ataxia. The recommended dose is 150 mg omaveloxolone (3 x 50 mg capsules) once daily.

SUMMARY:
Friedreich's ataxia (FA) is a rare, inherited neurodegenerative disease that typically begins in children and young people. It primarily affects the spinal cord, peripheral nerves and cerebellum of the brain. Clinical manifestations include progressive gait and limb ataxia, auditory and optic neuropathy, cardiomyopathy, scoliosis, dysarthria, and dysphagia. In advanced stages, individuals may become wheelchair-dependent, leading to a severe loss of autonomy and reduced life expectancy. To date, there are no effective treatments known to reverse or halt disease progression. Heart disease remains the leading cause of death in individuals with FA. In January 2024, Omaveloxolone was approved for early access in France to treat FA in patients aged 16 years and older. Dysphagia is a central manifestation in FA, and may lead to severe complications such as malnutrition, dehydration, and aspiration-related pneumonia, as well as reduced self-esteem and social isolation. Despite its clinical relevance, dysphagia remains underexplored in clinical trials, including in major Omaveloxolone studies where no specific tool for measuring dysphagia has been incorporated. This study aimed to comprehensively evaluate the effect of Omaveloxolone on dysphagia after six months of treatment, in a cohort of French patients with Friedreich's ataxia who benefited from early access to treatment between February 2024 and May 2025. The severity of dysphagia will be assessed using the Sydney Swallow Questionnaire (SSQ), completed by patients at baseline and after six months of Omaveloxolone treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 16 Years
* Confirmed diagnosis of Friedreich's ataxia, genetically verified.
* Omaveloxolone therapy between February 2024 and May 2025, having receive treatment for at least 6 months.

Exclusion Criteria:

* Participants who interrupted treatment permanently before 6 months.
* Participants who did not complete the SSQ (Sydney swallow Questionnaire) at baseline and after 6 months of treatment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be selected from two public hospitals in France Lille and Nice where patients with genetically confirmed Friedreich's ataxia were treated with early access Omaveloxolone treatment.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the progression of dysphagia after 6 months of treatment with Omaveloxolone. | At the time of treatment initiation and after 6 months of Omaveloxolone treatment
  The SARA (Scale for the Assessment and Rating of Ataxia) questionnaire has eight categories with accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia). Participants will be divided into three groups based on the SARA score. The analysis will compare the mean SSQ (Sydney Swallow Questionnaire) score within each group at the beginning of treatment and again after six months. Additionally, variations in SSQ scores across the three groups will be evaluated to identify any differences in the progression of dysphagia.

SECONDARY OUTCOMES:
Comparison between SSQ (Sydney Swallow Questionnaire) and SARA (Scale for the Assessment and Rating of Ataxia) scores | At the time of treatment initiation and after 6 months of Omaveloxolone treatment
  The SARA questionnaire has eight categories with accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia). Participants will be divided into three groups based on the SARA score. The analysis will compare the mean SSQ scores within each group at the beginning of treatment and again after six months. Additionally, variations in SSQ scores across the three groups will be evaluated to identify any differences in the progression of dysphagia.
Correlation after 6 months of treatment between SARA (Scale for the Assessment and Rating of Ataxia) and SSQ (Sydney Swallow Questionnaire) scores. | At the time of treatment initiation and after 6 months of Omaveloxolone treatment
  After 6 months of treatment, the correlation between neurological damage measured by SARA and dysphagia measured by SSQ will be evaluated.
Impact of functional status (ambulant vs. non-ambulant) on dysphagia | At the time of treatment initiation and after 6 months of Omaveloxolone treatment
  Participants will be divided into two groups: Ambulatory and Non-ambulatory and a comparison will be made between the SSQ (Sydney Swallow Questionnaire) scores at baseline and after six months within each group.
Correlation between GAA expansion size and dysphagia (SSQ score) Sydney Swallow Questionnaire | At the time of treatment initiation and after 6 months of Omaveloxolone treatment
  Participants will be divided into 3 groups based on the size of the GAA expansion on the shorter allele and SSQ scores .
Correlation between (GAA expansion) size GAA: a repeated sequence of three nucleotides: guanine (G), adenine (A), adenine (A) in DNA. and the evolution of neurological damage ( SARA score) Scale for the Assessment and Rating of Ataxia | At the time of treatment initiation and after 6 months of Omaveloxolone treatment
  The size of the GAA expansion is information that can be found in patients medical files. Participants will be divided into three groups based on the size of the GAA expansion and a comparison will be made between the ( SARA score) Scale

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, Alpes Maritimes, France